CLINICAL TRIAL: NCT03027128
Title: Open-label, Phase 1 Study of haNK™ for Infusion in Subjects With Metastatic or Locally Advanced Solid Tumors
Brief Title: QUILT-3.028: Study of haNK™ for Infusion in Subjects With Metastatic or Locally Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.028
Record Dates: First submitted 2017-01-18; First posted 2017-01-20 (Estimated); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: Solid Tumor
Keywords: Phase 1; Metastatic; Locally Advanced; Cancer; Cell Therapy
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort 1, 2x10^9 Cells haNK™ (Experimental): NK-92 [CD16.158V, ER IL-2], Suspension for Intravenous Infusion
  Interventions: Biological: haNK™ for Infusion

INTERVENTIONS:
Biological: haNK™ for Infusion — haNK™ for Infusion is a human, allogeneic, NK cell line that has been engineered to produce endogenous, intracellularly retained IL-2 and to express CD16, the high-affinity (158V) Fc gamma receptor (FcγRIIIa/CD16a).
  Other Names: NK-92 [CD16.158V, ER IL-2], Suspension for Intravenous

SUMMARY:
The purpose of this study is to determine whether haNK™ for Infusion is safe and effective in the treatment of metastatic or locally advanced solid tumors.

DETAILED DESCRIPTION:
This is a phase 1 trial in subjects with metastatic or locally advanced solid tumors. The study will be conducted in two parts: part 1 will involve dose escalation using a 3 + 3 design, and part 2 will involve the expansion of the MTD or HTD to further evaluate the safety of haNK. In part 1, 3 to 6 subjects will be sequentially enrolled starting at dose cohort 1, and subjects will be assessed for DLTs.

* Cohort 1: 2 x 10^9 cells per infusion.
* Cohort 2: 4 x 10^9 cells per infusion.
* If needed, subjects will be enrolled into a dose de-escalation cohort (cohort -1): 1 x 10^9 cells per infusion.

In part 2, dose expansion will occur when the MTD or HTD has been determined. An additional 4 subjects may be enrolled in part 2, for a total of up to 10 subjects at the MTD or HTD.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Able to understand and provide a signed informed consent that fulfills the relevant IRB or IEC guidelines.
3. Histologically confirmed, unresectable, locally advanced or metastatic solid malignancy.
4. ECOG performance status of 0 to 2.
5. Have at least 1 measurable lesion and/or non-measurable disease evaluable according to RECIST Version 1.1.
6. Must have a recent formalin-fixed, paraffin-embedded (FFPE) tumor biopsy specimen following the conclusion of the most recent anticancer treatment. If an historic specimen is not available, the subject must be willing to undergo a biopsy during the screening period, if considered safe by the Investigator. If safety concerns preclude collection of a biopsy during the screening period, a tumor biopsy specimen collected prior to the conclusion of the most recent anticancer treatment may be used.
7. Must be willing to provide pre- and post-infusion blood samples.
8. Have received treatment with at least 1 prior line of therapy in the metastatic setting or not be a candidate for therapy of proven efficacy for their disease. Prior immune therapy is allowed.
9. Resolution of all toxic side effects of prior chemotherapy, radiotherapy, or surgical procedures to CTCAE grade ≤ 1, with the exception of alopecia.
10. Life expectancy ≥ 12 weeks.
11. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
12. Agreement to practice effective contraception for female subjects of child-bearing potential and non-sterile males. Female subjects of child-bearing potential are considered all female subjects being physiologically capable of becoming pregnant. Female subjects of child-bearing potential are usually premenopausal women or women with less than 12 months of amenorrhea post-menopause and who have not undergone surgical sterilization. Female subjects of child-bearing potential and non-sterile male subjects must agree to use effective contraception for at least 60 days (female) and 120 days (male) after the last dose of haNK. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm) used with spermicide, intrauterine devices (IUDs), and abstinence.

Exclusion Criteria:

1. History of persistent grade 2 or higher (CTCAE Version 4.03) hematological toxicity resulting from previous therapy.
2. Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drug used in this study or that would put the subject at high risk for treatment-related complications.
3. Systemic autoimmune disease (eg, lupus erythematosus, rheumatoid arthritis, Addison's disease, autoimmune disease associated with lymphoma).
4. History of organ transplant requiring immunosuppression.
5. History of or active inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
6. Inadequate organ function, evidenced by the following laboratory results:

   * White blood cell (WBC) count < 2,500 cells/mm^3
   * Absolute neutrophil count < 1,500 cells/mm^3.
   * Platelet count < 100,000 cells/mm3.
   * Hemoglobin < 9 g/dL.
   * Total bilirubin greater than the upper limit of normal (ULN; unless the subject has documented Gilbert's syndrome).
   * Aspartate aminotransferase (AST [SGOT]) or alanine aminotransferase (ALT [SGPT]) > 2.5 × ULN (> 5 × ULN in subjects with liver metastases).
   * Alkaline phosphatase levels > 2.5 × ULN (> 5 × ULN in subjects with liver metastases, or >10 × ULN in subjects with bone metastases).
   * Serum creatinine > 2.0 mg/dL or 177 μmol/L.
7. Uncontrolled hypertension (systolic > 150 mm Hg and/or diastolic > 100 mm Hg) or clinically significant (ie, active) cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia requiring medication.
8. Dyspnea at rest due to complications of advanced malignancy or other disease requiring continuous oxygen therapy.
9. Positive results of screening test for human immunodeficiency virus (HIV). However, subjects with HIV are allowed on the study if they meet the following criteria:

   * CD4+ T-cell count >200 cells/mm^3.
   * Stable antiretrovital therapy for at least 12 weeks prior to entry.
   * Plasma HIV RNA levels below lower limit of quantification at screening, and no quantifiable HIV RNA levels within the 12 weeks preceding screening.
10. Current chronic daily treatment (continuous for > 3 months) with systemic corticosteroids (dose equivalent to or greater than 10 mg/day methylprednisolone), excluding inhaled steroids. Short-term steroid use to prevent IV contrast allergic reaction or anaphylaxis in subjects who have known contrast allergies is allowed.
11. Known hypersensitivity to any component of the study medication(s).
12. Participation in an investigational drug study or history of receiving any investigational treatment within 28 days prior to screening for this study, except for testosterone-lowering therapy in men with prostate cancer.
13. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
14. Concurrent participation in any interventional clinical trial.
15. Pregnant and nursing women. A negative serum pregnancy test within 72 hours before administration of haNK must be documented before any haNK is administered to a female subject of child-bear potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-05-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chan Soon-Shiong Institute for Medicine, El Segundo, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only Cohort 1 enrolled participants on this study.
Period: Overall Study
Arm/Group | Cohort 1, 2x10^9 Cells haNK™
Started | 6
Completed (Completed defined as receiving at least one dose of study drug.) | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cohort 1, 2x10^9 Cells haNK™
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Histology of Primary Diagnosis [Count of Participants; unit: Participants]
  Carcinoma/Adenocarcinoma | 4
  Epithelial | 1
  Squamous cell carcinoma | 1

OUTCOME MEASURES:

1. Primary Outcome: Determination of Maximum Tolerated Dose (MTD) or Highest Tested Dose (HTD).
Time Frame: 28 days/4 weeks
Population: All subjects that received at least one dose of study drug.
Measure: Number; unit: cells
Groups:
- Cohort 1: 2 x 10^9 Cells haNK™: NK-92 [CD16.158V, ER IL-2], Suspension for Intravenous Infusion
  haNK™ for Infusion: haNK™ for Infusion is a human, allogeneic, NK cell line that has been engineered to produce endogenous, intracellularly retained IL-2 and to express CD16, the high-affinity (158V) Fc gamma receptor (FcγRIIIa/CD16a).
Arm/Group | Cohort 1: 2 x 10^9 Cells haNK™
Number analyzed (Participants) | 6
cells | 2,000,000,000

2. Primary Outcome: Occurrence of Dose-limiting Toxicities (DLTs).
Time Frame: 28 days/4 weeks
Population: All subjects that received at least one dose of study drug.
Measure: Number; unit: Number of DLTs
Arm/Group | Cohort 1: 2 x 10^9 Cells haNK™
Number analyzed (Participants) | 6
Number of DLTs | 0

3. Primary Outcome: Number of Participants With Treatment-emergent Adverse Event (AEs) and Serious Adverse Events (SAEs)
Time Frame: The investigator will record all reportable events with start dates occurring any time after informed consent is obtained until 30 days after the last day of study participation, up to 5.3 months.
Population: All subjects that received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1: 2 x 10^9 Cells haNK™
Number analyzed (Participants) | 6
participants
  Treatment-emergent adverse event | 6
  Serious adverse events | 1

ADVERSE EVENTS:
Time Frame: The investigator will record all reportable events with start dates occurring any time after informed consent is obtained until 30 days after the last day of study participation, up to 5.3 months.
Arm/Group | Cohort 1: 2 x 10^9 Cells haNK™
All-Cause Mortality (participants affected / at risk) | 2/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 2 x 10^9 Cells haNK™ (N=6)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 2 x 10^9 Cells haNK™ (N=6)
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Fatigue (General disorders) | 5
Pyrexia (General disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2
Rib fracture (Injury, poisoning and procedural complications) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
There is an insufficient number of subjects enrolled in order to evaluate efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT03027128/Prot_SAP_000.pdf